CLINICAL TRIAL: NCT03368157
Title: PREG-MS: New England MS Pregnancy Prospective Cohort Study
Brief Title: PREG-MS: New England MS Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Maria Houtchens, Assistant Professor of Neurology, Brigham and Women's Hospital
Other Study IDs: 2016P000588
Record Dates: First submitted 2017-11-27; First posted 2017-12-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Pregnancy Related
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to develop a detailed pregnancy registry of patients with Multiple Sclerosis in the New England states. Women with a diagnosis of MS that are either pregnant or actively planning to become pregnant are eligible to participate.

The study will solely take place through phone interviews. One of the study coordinator at the Partners MS Center will contact the participant for an intake phone interview where general information about the individual, their pregnancy and their MS will be collected. Thereafter the coordinator will contact the participant every 3 months for 20 minutes follow up interviews. After birth, the coordinator will collect information on the growth and development of the participant's baby. Pediatric interviews will be conducted at 2, 4, 6, 9, 12, 18, 24, 36 months. Information from the participant's neurologist and obstetrician, as well as information from the baby's pediatrician, will be made available to the study staff at regular intervals throughout the duration of the study.

Through this study, the investigators hope to learn more about the effects of MS on pregnancy and pediatric development, and about the effects of pregnancy on the course of MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis;
* Pregnant or actively planning to become pregnant.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who are pregnant or are actively trying to become pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
The relationship between EDSS and pregnancy course | 9 months
  The investigators assessed the correlation between EDSS scores and the presence of pregnancy complications, or the lack thereof.

SECONDARY OUTCOMES:
The relationship between MS treatments and pregnancy course | 9 months
  The investigators assessed the effects of Disease modifying therapies used to treat MS and its implication on the pregnancy course.

OTHER OUTCOMES:
The weight (pounds) of infants born to MS affected mothers | 3 years
  The evaluation of the weight in pounds of infants born to mothers affected by MS compared to standard pediatric measurements.
The length (inches) of infants born to MS affected mothers | 3 years
  The evaluation of the length in inches of infants born to mothers affected by MS compared to pediatric standard measurements.
The head circumference (inches) of infants born to MS affected mothers | 3 years
  The evaluation of the head circumference in inches of infants born to mothers affected by MS compared to pediatric standard measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Houtchens MK, Manieri MC, Mahlanza TD, Pol-Patil J, Klawiter EC, Solomon AJ, Lathi E, Katz J, Ionete C, Morales IB, Severson C, Zurawski J, Stankiewicz JM, Cabot A, Sadovnick AD. A Real-World Prospective Multiple Sclerosis Pregnancy Registry in the United States: PREG-MS. Neurol Clin Pract. 2025 Apr;15(2):e200425. doi: 10.1212/CPJ.0000000000200425. Epub 2025 Jan 10. PMID 39810912